CLINICAL TRIAL: NCT06120933
Title: A Single-Group Clinical Trial Investigating the Effects of a Hair Vitamin Combination on Hair Growth and Hair Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrandiZone (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20354
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hair Health; Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test population (Experimental): For the first 8 weeks, each participant will take both the Hair Nutra Growth and Hair Nutra Boost supplements daily.
  For the remaining 4 weeks, participants will only take the Hair Nutra Growth supplement.
  Interventions: Dietary Supplement: Hair Nutra Growth Supplement & Hair Nutra Boost Supplement; Dietary Supplement: Hair Nutra Growth

INTERVENTIONS:
Dietary Supplement: Hair Nutra Growth Supplement & Hair Nutra Boost Supplement — Study Initiation (Week 0) to Week 8:
  Each participant will take both the Hair Nutra Growth capsules and the Hair Nutra Boost capsules.
  Participants should take 2 capsules of Hair Nutra Growth daily, one in the morning and one in the afternoon, with food or after a meal. The capsules should be taken with water.
  Participants should take 1 capsule of Hair Nutra Boost daily with food or after a meal. These capsules should also be taken with water.
Dietary Supplement: Hair Nutra Growth — From Week 9 to Week 12:
  Participants should ONLY take the Hair Nutra Growth. Participants should take 1 capsule of Hair Nutra Boost daily with food or after a meal. These capsules should also be taken with water.

SUMMARY:
This clinical trial aims to investigate the effectiveness of two Vitamins Revive hair supplements in promoting hair growth, reducing hair loss, and improving overall hair health. The products under assessment are Hair Nutra Growth and Hair Nutra Boost. The trial will assess the efficacy of the products to induce better hair growth, reduction in hair loss and shedding, increased hair thickness and fullness, and improvement in hair appearance and vitality over a 12-week testing period. Participants will complete study-specific questionnaires at Baseline, Week 4, Week 8, and Week 12. Participants will also provide photos of their hair at Baseline, Week 4, Week 8, and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Women Aged 30+ Self-reported issues with hair growth, shedding, and thinning Generally healthy - don't live with any uncontrolled chronic disease Must be willing to stop taking any other hair growth supplements or biotin supplements for the duration of the trial In the last three months, has not introduced any new supplements or medications to target hair growth, hair loss, or hair health Individuals must agree to refrain from dyeing their hair in the target interest areas until the study is complete Willing and able to take high-quality photographs of their hairline

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders Anyone with known severe allergic reactions Anyone with a known allergy to any of the ingredients Anyone currently using a hair growth supplement Anyone currently using biotin Anyone with scalp or hair diseases including but not limited to alopecia areata (a hair loss disorder leading to patchy bald spots on the head) Women who are pregnant, breastfeeding, or attempting to become pregnant Unwilling to follow the study protocol

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported rate of hair growth. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in self-reported rate of hair growth will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in self-reported rate of hair loss. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in rate of hair loss will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe"). Changes in self-reported rate of hair loss
Changes in hair shedding. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in hair shedding will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

SECONDARY OUTCOMES:
Changes in participant-percieved overall hair health. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in participants perception of their overall hair health will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

OTHER OUTCOMES:
Changes in hair thickness. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in participants' perception of their hair thickness will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in hair shine. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in participants' perception of their hair shine will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in hair softness. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in participants' perception of their hair softness will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in hair vitality. [Timeframe: Baseline to Week 12] | 12 weeks
  Changes in participants' perception of their hair vitality will be recorded via study-specific questionnaires. Responses will be on a Likert scale (0-5 scale), with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided